CLINICAL TRIAL: NCT02518633
Title: Assessment of Hypoxia in Adipose Tissue of Subjects With Obstructive Sleep Apnoea
Brief Title: Obstructive Sleep Apnoea and Adipose Tissue Dysfunction
Status: Completed | Type: Observational
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Principal Investigator, Katarina Kos, Consultant Physician, Royal Devon and Exeter NHS Foundation Trust
Other Study IDs: OSAadipose
Record Dates: First submitted 2015-03-23; First posted 2015-08-10 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Obstructive Sleep Apnoea; Obesity; Hypoxia
Keywords: obesity; hypoxia; adipose tissue
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity; Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — adipose tissue and blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- men with obstructive sleep apnoea: Continuous positive airway pressure devices
  Interventions: Device: Continuous positive airway pressure devices
- control subjects: subjects with no obstructive sleep apnoea

INTERVENTIONS:
Device: Continuous positive airway pressure devices — overnight use of CPAP device
  Other Names: CPAP
  Groups: men with obstructive sleep apnoea

SUMMARY:
Dysfunctional adipose tissue predisposes to cardiovascular disease. Similarly, the risk of cardiovascular disease appears to be increased in subjects with obstructive sleep apnoea. Reduced adipose tissue oxygen availability has been described in obesity and may also be a mechanism in obstructive sleep apnoea. Hypoxia induces inflammation and fibrosis in adipose tissue which are factors contributing to cardiovascular risk. The investigators hypothesize that adipose tissue's oxygen uptake is reduced in subjects with obstructive sleep apnoea by comparing in vivo AT oxygenation and blood flow in tissue of control subjects.

DETAILED DESCRIPTION:
Assessment includes a adipose tissue biopsy and measurement of oxygenation and blood flow by a Clarke type electrodes and non-invasive Doppler techniques.

ELIGIBILITY:
Inclusion Criteria:

* men with or without obstructive sleep apnoea

Exclusion Criteria:

* weight loss interventions
* steroid use
* active smoking

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with newly diagnosed obstructive sleep apnoea and controls
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-03; Primary Completion 2015-03 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
pO2 in adipose tissue by Clarke type electrode | 4 months
  Measurement of pO2 by Clarke type electrode

SECONDARY OUTCOMES:
blood flow in adipose tissue by laser Doppler techniques | 4 months
  assessment of tissue blood flow by laser Doppler techniques

OTHER OUTCOMES:
adipose tissue gene expression of HIF-1alpha | 4 months
  adipose tissue expression of hypoxia related genes

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Kos, FRCP,PhD, Principal Investigator — University of Exeter
Locations (2):
- United Kingdom (2):
  - NIHR Clinical Research Facility, Exeter
  - Royal Devon and Exeter NHS Foundation Trust, Exeter

REFERENCES:
- [Background] Thorn CE, Knight B, Pastel E, McCulloch LJ, Patel B, Shore AC, Kos K. Adipose tissue is influenced by hypoxia of obstructive sleep apnea syndrome independent of obesity. Diabetes Metab. 2017 Jun;43(3):240-247. doi: 10.1016/j.diabet.2016.12.002. Epub 2017 Jan 26. PMID 28131740